CLINICAL TRIAL: NCT02904265
Title: Non-inferiority Prospective Randomized Trial of Acetazolamide Versus Diazepam in Patients With Continuous Spike and Wave in Sleep (CSWS)/Landau Kleffner Syndrome (LKS)
Brief Title: Efficacy Study of Acetazolamide Versus Diazepam in Continuous Spike and Wave/Landau-Kleffner Syndrome
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Katherine C. Nickels, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-002442
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Landau-Kleffner Syndrome; Status Epilepticus, Electrographic
Keywords: continuous spike wave in sleep; Landau-Kleffner syndrome; acetazolamide; diazepam
MeSH Terms: conditions — Landau-Kleffner Syndrome; Status Epilepticus | interventions — Diazepam; Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diazepam (Active Comparator): Diazepam 0.5 mg/kg (up to maximum 20 mg) by mouth nightly. Duration of therapy is 4 weeks.
  Interventions: Drug: Diazepam
- Acetazolamide (Experimental): Acetazolamide 8-10 mg/kg (up to a maximum dose of 375 mg) by mouth (PO)divided twice daily X 1 week, then increased to 11-16 mg/kg (up to a maximum dose of 750 mg) by mouth divided twice daily thereafter. Duration of therapy is 4-8 weeks.
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Diazepam
  Other Names: Valium
  Arms: Diazepam
Drug: Acetazolamide
  Other Names: Diamox; Diamox Sequels
  Arms: Acetazolamide

SUMMARY:
The purpose of this study is to compare the effectiveness of the medications acetazolamide and diazepam in the treatment of continuous spike wave in sleep (CSWS) and Landau-Kleffner syndrome (LKS).

ELIGIBILITY:
Inclusion Criteria:

* ESES and clinical CSWS/LKS defined by all of the following:
* SWI ≥50% during first hour of sleep
* Bilateral synchrony of discharges during sleep
* Clinical evidence of behavior and/or academic regression
* Daytime SWI ≤20%

Exclusion Criteria:

* Previous treatment with benzodiazepine or acetazolamide for Electrical Status Epilepticus in Sleep (ESES)
* Current treatment with carbamazepine, phenytoin, oxcarbazepine, phenobarbital, vigabatrin or lamotrigine
* Antiepileptic medication changes over the month prior to enrollment
* Epileptic encephalopathy other than CSWS/LKS
* Prior serious adverse reaction to benzodiazepines or acetazolamide
* Sulfa allergy
* Progressive underlying neurologic condition
* Frequent seizures that would prevent the patient from maintaining a stable dose of medications
* Female patient that has begun menses or is pregnant

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2016-09; Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C. Nickels, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fine AL, Wirrell EC, Wong-Kisiel LC, Nickels KC. Acetazolamide for electrical status epilepticus in slow-wave sleep. Epilepsia. 2015 Sep;56(9):e134-8. doi: 10.1111/epi.13101. Epub 2015 Jul 31. PMID 26230617
- [Background] De Negri M, Baglietto MG, Battaglia FM, Gaggero R, Pessagno A, Recanati L. Treatment of electrical status epilepticus by short diazepam (DZP) cycles after DZP rectal bolus test. Brain Dev. 1995 Sep-Oct;17(5):330-3. doi: 10.1016/0387-7604(95)00076-n. PMID 8579219
- [Background] Francois D, Roberts J, Hess S, Probst L, Eksioglu Y. Medical management with diazepam for electrical status epilepticus during slow wave sleep in children. Pediatr Neurol. 2014 Mar;50(3):238-42. doi: 10.1016/j.pediatrneurol.2013.11.002. Epub 2013 Nov 12. PMID 24393416
- [Background] Katayama F, Miura H, Takanashi S. Long-term effectiveness and side effects of acetazolamide as an adjunct to other anticonvulsants in the treatment of refractory epilepsies. Brain Dev. 2002 Apr;24(3):150-4. doi: 10.1016/s0387-7604(02)00003-7. PMID 11934510
- [Background] Sanchez Fernandez I, Peters JM, An S, Bergin AM, Takeoka M, Rotenberg A, Kothare SV, Riviello JJ Jr, Loddenkemper T. Long-term response to high-dose diazepam treatment in continuous spikes and waves during sleep. Pediatr Neurol. 2013 Sep;49(3):163-170.e4. doi: 10.1016/j.pediatrneurol.2013.04.027. PMID 23953953
- [Background] Wirrell E, Ho AW, Hamiwka L. Sulthiame therapy for continuous spike and wave in slow-wave sleep. Pediatr Neurol. 2006 Sep;35(3):204-8. doi: 10.1016/j.pediatrneurol.2006.02.012. PMID 16939861
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study closed due to only 3 participants recruited
Pre-assignment Details: Study closed due to only 3 participants recruited
Groups:
- Diazepam: Diazepam 0.5 mg/kg (up to maximum 20 mg) by mouth nightly. Duration of therapy is 4 weeks.
  Diazepam
- Acetazolamide: Acetazolamide 8-10 mg/kg (up to a maximum dose of 375 mg) by mouth (PO)divided twice daily X 1 week, then increased to 11-16 mg/kg (up to a maximum dose of 750 mg) by mouth divided twice daily thereafter. Duration of therapy is 4-8 weeks.
  Acetazolamide
Period: Overall Study
Arm/Group | Diazepam | Acetazolamide
Started | 1 (Study closed due to only 3 participants recruited) | 2 (Study closed due to only 3 participants recruited)
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diazepam | Acetazolamide | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 1 | 2 [1 to 2] | 1.5 [1 to 3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Short-term Tolerability of Acetazolamide vs Diazepam
Description: Expect improved side effect profile of acetazolamide compared to diazepam at short-term follow up
Time Frame: 4-8 weeks of start of medications
Population: Study closed due to only 3 participants recruited
Measure: Count of Participants; unit: Participants
Arm/Group | Diazepam | Acetazolamide
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events will be assessed for the duration of the study for each subject, for approximately 6 months. All adverse events will be followed through to resolution or until the investigators attribute the adverse event to a cause other than the study drugs or assesses them as chronic or stable.
Description: Study was closed due to only 3 participants recruited
Arm/Group | Diazepam | Acetazolamide
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT02904265/Prot_SAP_000.pdf